CLINICAL TRIAL: NCT04810819
Title: Clinical Study of the Effect of Methylprednisolone Combined With Two Hydroxypropyl Theophylline on Respiratory Dynamics During Thoracoscopic Lobectomy
Brief Title: Clinical Study of the Effect of Methylprednisolone Combined
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: contrast-2021
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Methylprednisolone;Dihydroxypropyltheophylline;One Lung Ventilation;Respiratory Dynamics
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Methylprednisolone 40 MG Injection;Dihydroxypropyltheophylline;
- control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone 40 MG Injection;Dihydroxypropyltheophylline; — Before anesthesia induction, 80 mg methylprednisolone and 100 ml saline were given intravenously, and 0.25 g dihydroxypropyltheophylline and 100 ml normal saline were given intravenously.
  Arms: Experimental group
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
Through the design of RCT study, the preoperative use of drugs (methylprednisolone + dihydroxypropyltheophylline) as intervention measures, the patients undergoing thoracoscopic lobectomy as the main research object, through the comparison of two groups of patients with intraoperative respiratory dynamics index and postoperative complications, to explore a more effective perioperative management method.

ELIGIBILITY:
Inclusion Criteria:

* 1. After fully understanding the purpose and significance of the trial, the patients voluntarily participated in the trial and signed the informed consent;

  2. The type of operation was general anesthesia and thoracoscopic lobectomy;

  3. Age 18-75 years old, including boundary value, gender is not limited;

  4. BMI 18-26kg / m2;

  5. ASA grade I-II; no mental disorder, normal consciousness, normal communication;

  6. No contraindications of methylprednisolone and dihydroxypropyltheophylline.

Exclusion Criteria:

* 1. There were diseases of immune, endocrine, nervous and mental system before operation, and serious dysfunction of heart, liver and kidney;

  2. Take immunosuppressive drugs and non steroidal anti-inflammatory drugs before operation;

  3. Respiratory tract infection (cough, expectoration, suffocation, etc.) in recent 1 month; pneumonia, bronchitis, etc. on CT;

  4. History of chronic pulmonary disease, including but not limited to asthma, pulmonary abscess, tuberculosis, chronic bronchitis, etc;

  5. FEV1 < 50%;

  6. Oxygen saturation was lower than 90% and airway pressure was higher than 40 cm H20;

  7. Continuous hypotension or hypertension during the operation; intraoperative blood loss > 1000ml;

  8. Allergic to methylprednisolone or dihydroxypropyltheophylline;

  9. There are any other situations that the researchers think are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Pplat | 5 different time points during the operation
  Airway pressure at different time points during operation
Ppeak | 5 different time points during the operation
  Peak airway pressure at different time points during operation